CLINICAL TRIAL: NCT05418413
Title: Dentoskeletal Changes Resulting From Treatment of Skeletal Class II With an Esthetic Twin Block Appliance.
Brief Title: The Use of an Esthetic Twin Block for Patients With Mandibular Retrusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-12-2022
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Class II Malocclusion
Keywords: Class II; Twin Block; Functional Therapy
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Twin-block appliance (Active Comparator): The patients in this control group will be treated using the conventional Twin-block appliance (CTB).
  Interventions: Device: CTB
- Esthetic Twin-block appliance (Experimental): the patients in this experimental group will be treated using the esthetic Twin-block appliance (ETB).
  Interventions: Device: ETB

INTERVENTIONS:
Device: CTB — conventional Twin-block (CTB) will be comprised of maxillary and mandibular removable appliances having the labial bows, adam's clasps, and with no incisal capping.
  Arms: Conventional Twin-block appliance
Device: ETB — will be comprised of maxillary and mandibular removable 1.5-mm biocryl sheet will be adapted separately on maxillary and mandibular casts with help of vacuum machine, and Acrylic bite blocks with the inclined plane will be fabricated on biocryl sheets sim
  Arms: Esthetic Twin-block appliance

SUMMARY:
This experimental study will evaluate the effect of an esthetic Twin-block appliance on the correction of class II malocclusion compared with the traditional Twin-block appliance.

The study sample will consist of 50 patients with class II malocclusion. The sample will be allocated randomly into two groups: the control group and the experimental group.

The traditional Twin-block appliance will be applied for the control group patients, while the esthetic Twin-block appliance will be applied for the experimental group patients. The dentoskeletal, soft tissue changes and esthetic and functional efficacy occurring after functional treatment will be assessed using cephalometric radiographs and profile photographs, pre and post-treatment, and a questionnaire. Changes for each group will be evaluated individually, and the two groups will be compared.

DETAILED DESCRIPTION:
Class II malocclusion is one of the most frequent orthodontic problems, and most class II malocclusion cases are the result of mandibular deficiency. Twin block (TB) is one of the most popular functional appliances to treat this condition. Despite excellent treatment results with TB, its acceptance and compliance may be hampered by its wiry structure and appearance. Furthermore, it has a side effect of causing the proclination of lower incisors, which reduces skeletal change. Various modifications were proposed to reduce lower incisors proclination but had no significant effect. Patient cooperation is one of the most important factors for successful functional appliance treatment, and it depends upon comfort and esthetic acceptability, which ensures good patient compliance. so, in order to enhance the esthetic appearance and overcome the disadvantages of a conventional Twin-Block (CTB), a novel esthetic Twin-Block (ETB) was fabricated from a specific material using a pressure molding device and acrylic bite blocks. There is only one study that evaluated this appliance which is a pilot study that compared the treatment effects of the (ETB) and (CTB) in the treatment of Class II malocclusions. However, this study has a lot of limitations, making it difficult to evaluate this appliance's efficiency accurately. The aim of this study is to study the dento-skeletal, soft tissue changes, and esthetic and functional efficacy that result from treatment by this appliance (ETB) and to compare them to the changes in the matched group will be treated with (CTB), by studying the cephalometric radiographs, profile photographs, and a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Angle class II malocclusion because of mandibular retrognathia
* O.J > 5 , SNB < 78
* Patient during growth spurt
* Normal or horizontal growth pattern Björk > 402

Exclusion Criteria:

* TMJ disorders
* Poor oral hygiene
* Previous orthodontic treatment.
* Patients with syndromes, clefts, or craniofacial abnormalities.
* Reason of contraindication of functional treatment

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Dentoskeletal mandible changes as measured by tomographic | Assessment will be done before treatment (T0) and after obtaining 0-1.5 mm overjet and the occlusion settled into a class I or superclass I molar relationship which will be approximately obtained after 8 months (T1).
  changes of the mandible before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs
Lower incisor angle changes | Changes will be evaluated before treatment and after obtaining 0-1.5 mm overjet and the occlusion settled into a class I or superclass I molar relationship which will be approximately obtained after 8 months (T1)
  Lower incisor angle changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.
ANB angle changes | Changes will be evaluated before treatment and after obtaining 0-1.5 mm overjet and the occlusion settled into a class I or superclass I molar relationship which will be approximately obtained after 8 months (T1)
  ANB angle changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.

SECONDARY OUTCOMES:
Dentoskeletal maxilla changes as measured by tomographic superimposition of the cranial base | Assessment will be done before treatment (T0) and after obtaining 0-1.5 mm overjet and the occlusion settled into a class I or superclass I molar relationship which will be approximately obtained after 8 months (T1)
  changes of the maxilla before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.
SNA angle changes | Assessment will be done before treatment (T0) and after obtaining 0-1.5 mm overjet and the occlusion settled into a class I or superclass I molar relationship which will be approximately obtained after 8 months (T1)
  SNA angle changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.
SNB angle changes | Assessment will be done before treatment (T0) and after obtaining 0-1.5 mm overjet and the occlusion settled into a class I or superclass I molar relationship which will be approximately obtained after 8 months (T1).
  SNB angle changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.
Soft tissue changes | Assessment will be done before treatment (T0) and after obtaining 0-1.5 mm overjet and the occlusion settled into a class I or superclass I molar relationship which will be approximately obtained after 8 months (T1)
  Soft tissue changes before and after treatment will be assessed and compared with those of the control group (Facial convexity angle, Nasolabial angle, Z-Merrifield angle, …etc) using profile photography.
The duration of functional treatment | After obtaining 0-1.5 mm overjet and the occlusion settled into a class I or superclass I molar relationship which will be approximately obtained after 8 months
  The duration of the functional treatment will be measured and compared between groups.
Levels of pain | A questionnaire will be given to the patients five times during treatment; after 1 week, after 1 week, after 6 weeks, after 3 months and at the end of the application of the appliance.
  The level of pain will be assessed and compared with those of the control group using a questionnaire with a Visual Analog Scale (VAS). The VAS is a 10-cm horizontal line with two focal points at its beginning and end (0: there is no pain - 10: the worst pain).
Levels of discomfort | A questionnaire will be given to the patients four times during treatment; after 1day, after 1 week, after 6 weeks, after 3 months and at the end of the application of the appliance.
  The level of discomfort will be assessed and compared with those of the control group using a questionnaire with a Visual Analog Scale (VAS). The VAS is a 10-cm horizontal line with two focal points at its beginning and end (0: there is no discomfort - 10: the worst discomfort).
Levels of acceptance | A questionnaire will be given to the patients four times during treatment; after 1day, after 1 week, after 6 weeks, after 3 months and at the end of the application of the appliance.
  The level of acceptance will be assessed and compared with those of the control group using a questionnaire with a Visual Analog Scale (VAS). The VAS is a 10-cm horizontal line with two focal points at its beginning and end (0: no acceptance - 10: the best acceptance).
Number of broken appliances | During the treatment time which will take approximately 8 months.
  The number of broken will be counted and compared with those of the control group .

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Najati Alsilq, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohamed Youssef, DDS,MSc,PhD, Study Director — Professor of Orthodontics, University of Damascus, Dental School, Damascus, Syria.
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sidlauskas A. Clinical effectiveness of the Twin block appliance in the treatment of Class II Division 1 malocclusion. Stomatologija. 2005;7(1):7-10. PMID 16254470
- [Background] Tripathi T, Singh N, Rai P, Gupta P. Comparison of Dentoskeletal Changes, Esthetic, and Functional Efficacy of Conventional and Novel Esthetic Twin Block Appliances among Class II Growing Patients: A Pilot Study. Turk J Orthod. 2020 Jun 1;33(2):77-84. doi: 10.5152/TurkJOrthod.2020.19030. eCollection 2020 Jun. PMID 32637187
- [Background] Baccetti T, Franchi L, Toth LR, McNamara JA Jr. Treatment timing for Twin-block therapy. Am J Orthod Dentofacial Orthop. 2000 Aug;118(2):159-70. doi: 10.1067/mod.2000.105571. PMID 10935956
- [Background] Shahamfar M, Atashi MHA, Azima N. Soft Tissue Esthetic Changes Following a Modified Twin Block Appliance Therapy: A Prospective Study. Int J Clin Pediatr Dent. 2020 May-Jun;13(3):255-260. doi: 10.5005/jp-journals-10005-1759. PMID 32904097
- [Background] van der Plas MC, Janssen KI, Pandis N, Livas C. Twin Block appliance with acrylic capping does not have a significant inhibitory effect on lower incisor proclination. Angle Orthod. 2017 Jul;87(4):513-518. doi: 10.2319/102916-779.1. Epub 2017 Jan 27. PMID 28128634
- [Derived] Alsilq MN, Youssef M. Soft tissue effects of aesthetic and conventional twin block appliances in the treatment of skeletal class II malocclusion: a randomized controlled trial. Sci Rep. 2025 Oct 28;15(1):37627. doi: 10.1038/s41598-025-21538-w. PMID 41152368
- [Derived] Alsilq MN, Youssef M. Dentoskeletal effects of aesthetic and conventional twin block appliances in the treatment of skeletal class II malocclusion: a randomized controlled trial. Sci Rep. 2025 Jan 13;15(1):1879. doi: 10.1038/s41598-025-86219-0. PMID 39805909